CLINICAL TRIAL: NCT04447456
Title: Comparison of Voice Results at 5 Years of Treatment of Glottic Squamous Cell Carcinoma T1 by Surgery Versus Radiotherapy
Acronym: VO Qual
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_68; 2020-A00738-31 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Glottic Carcinoma
Keywords: Glottic Squamous Cell Carcinoma; Surgery; Radiotherapy; Voice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery
- Radiotherapy

SUMMARY:
Patients with early-stage squamous cell carcinomas of the vocal cord can be treated in an equivalent way in terms of carcinology by surgery or radiotherapy. The study will be to analyse the vocal outcome at 5 years of these two types of management in order to define whether one is superior to the other on this criterion of voice quality after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glottic squamous cell carcinoma T1N0M0 who may benefit from treatment with exclusive radiotherapy or exclusive surgery.
* patients treated for these cancers at Lille University Hospital and the Oscar Lambret Centre between 2015 and 2017.
* Tis, T1a and T1b glottic squamous cell carcinomas according to the TNM 7th edition classification in long-term survivors.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated for glottic squamous cell carcinoma at Lille University Hospital and the Oscar Lambret Centre between 2015 and 2017.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index | At 5 years
  The VHI is a self-administered questionnaire that provides a score ranging from 0 to 120 points validated in France and internationally based on the declarative answers to 30 items of the questionnaire. A high score corresponds to a voice felt to be of poor quality. This is a subjective assessment made by the patient.

SECONDARY OUTCOMES:
Maximum Phonation Time | At 5 years
  The TMP is the measurement in seconds of a vowel (/a/) held for as long as possible.
Grade, Roughness, Breathiness, Asthenia, Strain, Instability SCORE (GRBASI Score) | At 5 years
  This score is obtained from an internationally and nationally validated hetero-assessment. It consists in the attribution by a listening jury made up of two people of a mark ranging from 0 to 3 for each of the 6 items: Grade, Roughness, Breathiness, Asthenia, Strain, Instability.
  A high score is associated with a voice perceived as bad by the audience.
Acoustic Analysis by Vocalab software | At 5 years
  short recording of the patient's voice delivering a standardized speech on VOCALAB software validated by the scientific community.

CONTACTS AND LOCATIONS:
Overall Officials: François Mouawad, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - Hôpital Huriez, CHU, Lille

REFERENCES:
- [Derived] Louison J, Labreuche J, Liem X, Rysman B, Morisse M, Mortuaire G, Mouawad F. Voice quality after surgery or radiotherapy for glottic T1 squamous cell carcinoma: Results of the VOQUAL study. Cancer Radiother. 2024 Aug;28(4):373-379. doi: 10.1016/j.canrad.2024.03.004. Epub 2024 Aug 9. PMID 39122636